CLINICAL TRIAL: NCT04427371
Title: Zhongda Hospital, School of Medicine, Southeast University
Brief Title: The Effect and Mechanism of lncRNA NBR2 Regulating Endothelial Pyroptosis by Targeting GSDMD in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Dr., Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: SoutheastUChina
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Sepsis
Keywords: endothelial cell injury; pyroptosis; lncRNA NBR2; gasdermin D
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survivors: Improve or under treatment
  Interventions: Other: the levels of pyroptosis
- nonsurvivors: all-cause 28-day mortality
  Interventions: Other: the levels of pyroptosis

INTERVENTIONS:
Other: the levels of pyroptosis — Blood samples were taken to detect plasma lncRNA NBR2 levels and GSDMD protein level.

SUMMARY:
Sepsis is a life-threatening disease characterized by multi-organ failure due to dysregulated host response to infection, with high global mortality of 30-50%. One of the most important pathophysiologic hallmarks in sepsis is vascular endothelial injury that contributes to the severity and outcome of the syndrome. Effective treatments for endothelial cell injury in sepsis have been lacking to improve prognosis. Endothelial pyroptosis is a vital mechanism of vascular endothelial injury in sepsis; mitigation or abolishment of endothelial cell pyroptosis alleviate vascular endothelial damage and improve the prognosis of sepsis mice. Gasdermin D (GSDMD) mediated endothelial pyroptosis plays a critical role in modulating vascular endothelial injury in sepsis.

Long non-coding RNA (lncRNA), as a class of non-coding protein RNA longer than 200 kD, contributes to a variety of cell biological processes. The dysregulation of lncRNA results in the occurrence and development of tumors, diabetes, sepsis and other diseases. Therefore, we detected lncRNA and mRNA expression profile in 26 blood samples of septic patients using Arraystar LncRNA Microarray. We found lncRNA NBR2 regulates septic endothelial pyroptosis.

To assess any correlation of pyroptosis levels with relevant endothelial cell injury parameters and determine the prognostic value in septic patients. we measured the levels of pyroptosis in patients admitted to the Department of Critical Care Medicine for sepsis and investigated the correlation with related markers of endothelium injury. Furthermore, we determined the prognostic value of pyroptosis levels for the mortality of patients with sepsis.

DETAILED DESCRIPTION:
We measured the levels of pyroptosis in patients admitted to the Department of Critical Care Medicine for sepsis and investigated the correlation with related markers of endothelium injury. Furthermore, we determined the prognostic value of pyroptosis levels for the mortality of patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed infection
* The sequential organ failure score (SOFA score) increases by more than or equal to 2 points on the basis
* Sign the informed consent

Exclusion Criteria:

1. the age < 18 or > 80 years of age
2. pregnant
3. tumor
4. viral hepatitis or liver cirrhosis
5. chronic renal tubular nephritis, chronic renal insufficiency
6. ulcerative colitis or crohn's disease
7. active systemic lupus erythematosus (SLE)
8. acute myocardial infarction
9. acute pancreatitis
10. engaged in other clinical subjects

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: sepsis was defined according to "sepsis 3.0", which including suspected or confirmed infection and increased SOFA ≥ 2, confirmed by two experienced intensive care physicians. The infection was defined on the basis of infection sites, clinical features, clinical microbiology, and imaging tests. Septic shock was defined as a vasopressor requirement to maintain a mean arterial pressure of 65 mmHg or greater and serum lactate level greater than 2 mmol/L in the absence of hypovolemia.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28-day
  all-cause 28-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No